CLINICAL TRIAL: NCT03166774
Title: Support of the Sexual Health in Oncology
Status: Withdrawn | Type: Observational
Why Stopped: The study stopped because the the project was abandoned.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: AssO
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Oncology; Sexual Health
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient consulting in oncology ervice: Program of support of the sexual health in oncology by questionnaire
  Interventions: Other: Program of support of the sexual health

INTERVENTIONS:
Other: Program of support of the sexual health — Patients included in the study have to answer to a questionnaire

SUMMARY:
Implementation of sexual health support program in oncology department. This program is organized in 3 axes. One is to inform the side effects of treatment on sexual health.

There is a counselling team (nurse, esthetician,sexologue..etc) to raise the subject with patient and partner .

Finally, the oncologist continue during the treatment to evaluate the benefit of this program and adapt their counselling according to the needs

ELIGIBILITY:
Inclusion Criteria:

* all patient consulting in oncology service
* age > 18 years
* accepting to participate

Exclusion Criteria:

* Age< 18 years
* Refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient followed in oncology
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Estimated)

PRIMARY OUTCOMES:
Benefit of the care measurement program | Day 1
  assessment of data recorded on questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra SCHULTZ, Psychologist, Principal Investigator — Fondation Hôpital Saint-Joseph

IPD SHARING:
Plan to Share IPD: No